CLINICAL TRIAL: NCT04833803
Title: Development of the Eating Behaviour Lapse Inventory Survey Singapore (eBLISS):An Exploratory Mixed-method Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National University Health System, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Principal Investigator, Jocelyn Chew, Research Fellow, National University Health System, Singapore
Other Study IDs: 2020/01439
Record Dates: First submitted 2021-04-05; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Eating Behavior
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: eBLISS — a novel instrument -Eating Behaviour Lapse Inventory Survey Singapore (eBLISS)- will be developed

SUMMARY:
An exploratory mixed-method study will be conducted to develop an instrument for early detection and prevention of overconsumption.

ELIGIBILITY:
Inclusion Criteria:

1. Above the legal age of 21 years old
2. Have a BMI ≥ 23kg/m2
3. Able to understand and read English language
4. Uses a smart phone that can download apps
5. Able to provide informed consent

Exclusion Criteria:

1. Diagnosed with a pre-existing psychological disorder such as anxiety and depression except binge eating disorder
2. Participating in a concurrent weight management intervention that is beside the usual care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are overweight or obese and are following up at the Centre for Obesity Management and Surgery (COMS) at the National University Hospital (NUH).
Sampling Method: Non-Probability Sample
Enrollment: 530 (Estimated)
Dates: Start 2021-04-12 (Estimated); Primary Completion 2023-03-22 (Estimated); Study Completion 2023-03-22 (Estimated)

PRIMARY OUTCOMES:
Self-regulation of Eating Behaviour Questionnaire (SREBQ) | 2021-2023

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chew HSJ, Chew NW, Loong SSE, Lim SL, Tam WSW, Chin YH, Chao AM, Dimitriadis GK, Gao Y, So JBY, Shabbir A, Ngiam KY. Effectiveness of an Artificial Intelligence-Assisted App for Improving Eating Behaviors: Mixed Methods Evaluation. J Med Internet Res. 2024 May 7;26:e46036. doi: 10.2196/46036. PMID 38713909
- [Derived] Chew HSJ, Lim SL, Kim G, Kayambu G, So BYJ, Shabbir A, Gao Y. Essential elements of weight loss apps for a multi-ethnic population with high BMI: a qualitative study with practical recommendations. Transl Behav Med. 2023 Apr 3;13(3):140-148. doi: 10.1093/tbm/ibac090. PMID 36689306